CLINICAL TRIAL: NCT04747197
Title: A Phase 1, Multicenter, Prospective, Open-Label, Dose Escalation Study of EYP-1901, a Tyrosine Kinase Inhibitor (TKI), in Subjects With Wet AMD
Brief Title: First in Human Study to Evaluate the Safety and Tolerability of EYP-1901 in Patients With Wet Age Related Macular Degeneration (wAMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EYP-1901-001
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: wAMD; EYP-1901; EyePoint; DAVIO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 440 ug, single dose (Experimental): EYP-1901 440 ug, single dose
  Interventions: Drug: EYP-1901
- 2060 ug, single dose (Experimental): EYP-1901 2060 ug, single dose
  Interventions: Drug: EYP-1901
- 3090 ug, single dose (Experimental): EYP-1901 3090 ug, single dose
  Interventions: Drug: EYP-1901

INTERVENTIONS:
Drug: EYP-1901 — Intravitreal injection

SUMMARY:
Phase 1 open-label study to assess the bioactivity, ocular and systemic safety, tolerability, and pharmacokinetics of a single dose injections of EYP-1901 at three dose levels: 440 µg, 2060 µg and 3090 µg in subjects with Wet Age Related Macular Degeneration (wAMD)

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with wet Age-Related Macular Degeneration (wAMD), in the study eye.
* Subject must have received ≥3 prior injections with the same anti-VEGF product: bevacizumab, ranibizumab, or aflibercept) in the 6 months prior to the Screening Visit, in the study eye.
* Demonstrated response to the intravitreal anti-vascular endothelial growth factor (VEGF) treatment in the study eye.
* Best-corrected visual acuity (BCVA) using ETDRS charts of 25 letters (20/320 Snellen equivalent) to 85 letters (20/20 Snellen equivalent).

Exclusion Criteria:

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye.
* Subfoveal fibrosis or scarring >50% of the total lesion, or atrophy in the study eye, confirmed by central reading center.
* Choroidal neovascularization (CNV) in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia that would compromise vision in the study eye, confirmed by central reading center.
* Any concurrent intraocular condition in the study eye (e.g., cataract or glaucoma) that, in the opinion of the Investigator, would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of the study results.
* Active intraocular inflammation (grade trace or above) in the study eye.
* History of rhegmatogenous retinal detachment or treatment for retinal detachment or macular hole (stage 3 or 4) in the study eye.
* History of idiopathic or autoimmune-associated uveitis in either eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular (study eye) and systemic treatment emergent adverse events (TEAEs) | Week 48
  Number of ocular (study eye) and systemic TEAEs during the treatment period - Intent-to-Treat (ITT) Population

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) by EDTRS | Baseline, Week 48
  Mean change from Baseline in BCVA in the Study Eye
Mean change in central subfield thickness (CST) | Baseline, Week 48
  Mean change from Baseline in CST measured in microns by Spectral-domain - optical coherence tomography (OCT) assessments by a study-certified OCT technician in the study eye

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - EyePoint Investigational Site, Phoenix, Arizona
  - EyePoint Investigational Site, Beverly Hills, California
  - EyePoint Investigative Site, Mountain View, California
  - EyePoint Investigational Site, Oxnard, California
  - EyePoint Investigational Site, Melbourne, Florida
  - EyePoint Investigational Site, St. Petersburg, Florida
  - EyePoint Investigational Site, Springfield, Massachusetts
  - EyePoint Investigative Site, Asheville, North Carolina
  - EyePoint Investigational Site, Philadelphia, Pennsylvania
  - EyePoint Investigational Site, Abilene, Texas
  - EyePoint Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel S, Storey PP, Barakat MR, Hershberger V, Bridges WZ Jr, Eichenbaum DA, Lally DR, Boyer DS, Bakri SJ, Roy M, Paggiarino DA. Phase I DAVIO Trial: EYP-1901 Bioerodible, Sustained-Delivery Vorolanib Insert in Patients With Wet Age-Related Macular Degeneration. Ophthalmol Sci. 2024 Apr 9;4(5):100527. doi: 10.1016/j.xops.2024.100527. eCollection 2024 Sep-Oct. PMID 38881599